CLINICAL TRIAL: NCT04844801
Title: Comparison of Three Care Strategies in Cases of New-onset Supraventricular Arrhythmia During Septic Shock : a Randomized Controlled Trial
Brief Title: Rate, Rhythm or Risk Control for New-onset Supraventricular Arrhythmia During Septic Shock: a Randomized Controlled Trial
Acronym: CAFS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: APHP190070
Record Dates: First submitted 2021-02-26; First posted 2021-04-14 (Actual); Last update posted 2026-01-07 (Actual); Status verified 2026-01

CONDITIONS: Supraventricular Arrhythmia; Septic Shock
Keywords: New-onset supraventricular arrhythmia; Atrial fibrillation; Septic shock; Critically ill patient; Strategies; Antiarrhythmic drugs
MeSH Terms: conditions — Shock, Septic; Atrial Fibrillation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Risk control strategy (Active Comparator): Magnesium sulfate + control of the modifiable NOSVA risk factors
  Interventions: Procedure: Risk control strategy
- Heart-Rate control strategy (Active Comparator): Risk-control + "low-dose" amiodarone
  Interventions: Procedure: Heart-Rate control strategy:
- Rhythm control strategy (Active Comparator): Risk-control + "high-dose" amiodarone +/- electrical cardioversion
  Interventions: Procedure: Rhythm control strategy:

INTERVENTIONS:
Procedure: Risk control strategy — * Magnesium sulfate 2g intravenous bolus over 20 mn (if creatinine clearance >30 mL/min)
  * Control of the modifiable NOSVA risk factors: hypovolemia, sepsis, metabolic disorders (e.g., hypokalemia, hyponatremia), acidosis, hypoxia, excess cardiac inotropism of vasopressors, central venous catheter malposition, hyperthermia.
  Arms: Risk control strategy
Procedure: Heart-Rate control strategy: — * Risk-control as described above
  * "Low dose" amiodarone:
    * Intravenous loading bolus (day-1): bolus of 4 mg/kg IV over 1hour (maximum 300 mg IV over 1 hour )
    * Enteral maintenance dose (oral or via gastric tube) (day-1 to day-7) 200mg/24hour in a single dose for 7 days (150 mg intravenous over 1hour if enteral route is unavailable)
  Arms: Heart-Rate control strategy
Procedure: Rhythm control strategy: — * Risk control as described above
  * "High dose" amiodarone:
    * Intravenous loading dose (day-1): initial bolus 7 mg/kg over 1 hour (maximum 600 mg i.e. 4 IVL vials over 1 hour); followed by continuous intravenous maintenance: for a total of 1200 mg over the first 24 hours (infusion pump)
    * Enteral dose maintenance Day-2 and day-3: 1200 mg/ 24 hours in three doses for 48hours (720 mg continuous intravenous over 24 hours if enteral route is unavailable).
  Day-4 to day-7: 200 mg/24 hours once a day (150 mg intravenous over 1hourr if enteral route is unavailable) - Electrical cardioversion (only in patients intubated on mechanical ventilation)
  1 to 3 external electric shocks starting at 200J if:
  * NOSVA persists after initial bolus of amiodarone AND norepinephrine base (or epinephrine base) doses > 0.3 µg/kg/min;
  * NOSVA persists more than 6 hours after initial IV loading dose of amiodarone. NB: Beyond day 7 (or after discharge from intensive care if this occurs before da
  Arms: Rhythm control strategy

SUMMARY:
New-onset supraventricular arrhythmia (NOSVA) is reported in 40 % of patients with septic shock and is associated with hemodynamic alterations and mortality. The lack of consensus regarding best practices for the management of NOSVA in this setting has led to major variations in practice patterns. Observational studies reported three usual strategies: (i) heart rate control (hereafter rate control) with the use of antiarrhythmic drugs, essentially based on low dose of amiodarone, (ii) rhythm control with the use of antiarrhythmic drugs, essentially based on high dose of amiodarone, and electrical cardioversionand (iii) modifiable NOSVA risk factors control (hereafter risk control) without using antiarrhythmic drugs.

Risk control would minimize adverse events of antiarrhythmic drugs. Rhythm control would rapidly improve haemodynamics via restoring diastole and decreasing cardiac metabolic demand, while minimizing exposure to anticoagulation. Heart-Rate control, would limit potential adverse events of high dose of amiodarone and of electrical cardioversion (only in patients intubated on mechanical ventilation), while controlling haemodynamics. Therefore, it seems important to compare these three strategies.

Our hypothesis is dual: first, that heart-rate control and rhythm control each improve hemodynamics with in fine a decreased mortality, as compared to a risk control; second, that rhythm control outperforms rate control in this setting.

This is a multicenter, parallel-group, open-label, randomized controlled superiority trial to compare the effectiveness and safety of these three strategies (risk control, rate control and rhythm control) for NOSVA during septic shock.

DETAILED DESCRIPTION:
All consecutive adult patients admitted to the intensive care unit with NOSVA during septic shock will be included in the presence of inclusion criteria and in the absence of exclusion criteria.

Randomization, performed immediately after the inclusion (Day-1), in 1:1:1 ratio will be stratified on center. Then the patient will receive the randomized strategy: risk control, rate control or rhythm control.

Before inclusion, the informed consent will be proposed to the patient. If the patient is unable to give his/her consent, the informed consent of the next-of-kin will be sought by study investigator. In the case the next-of-kins are unidentified and/or unreachable, an emergency procedure will be applied. Patient consent will be sought as soon as their state of health allows it.

According to clinical guidelines, patients in all groups will receive therapeutic anticoagulation if NOSVA > 48 hours and in the absence of contraindication. In all groups, recommendations for the management of septic shock will be followed.

After day-7 (or hospital discharge if before J7), NOSVA treatment will be left at the discretion of attending physicians.

Evaluation criteria will be collected at day-2, day-3, day-7 (or at hospital discharge if before day-7), at the day of ICU discharge and at Day-28. If the patient has been discharged before Day-28, the vital status may be obtained by phone call at Day-28.

ELIGIBILITY:
Inclusion Criteria:

1. Age >= 18 years
2. Septic shock, defined by the association of the following criteria:

   * Documented or suspected infection, with initiation of antibiotic therapy
   * Initiation of vasopressors (norepinephrine, epinephrine) for at least 1 hour to maintain the MAP > 65 mmHg
3. NOSVA with heart rate ≥ 110 bpm lasting 5 minutes or more
4. Written informed consent (patient, next of skin or emergency situation)
5. Affiliation to a social security system

Exclusion Criteria :

1. Refractory shock defined by a dose of noradrenaline BASE or adrenaline BASE > 1.2 µg/kg/min
2. Cardiac surgery or cardiac transplant in the previous month
3. Aortic or mitral mechanical prosthesis, significant mitral stenosis (mitral surface < 1.5 cm2)
4. Congenital heart disease other than bicuspid aortic valve, atrial defect or patent foramen ovale.
5. History of supraventricular arrhythmia prior to the episode of septic shock defined by a permanent TRSVN or paroxysmal TRSVN requiring long-term specific treatment (heart rate reducer and/or antiarrhythmic and/or curative anticoagulation) or permanent NOSVA.
6. NOSVA that began more than 48 hours ago * (or more than 24 hours ago under vasopressor). * In cases of TRSVN dating back more than 48 hours, the patient may be included after undergoing a transesophageal echocardiogram (only in patients who are intubated and on mechanical ventilation) to rule out the presence of an intracardiac thrombus, coupled with the initiation of curative anticoagulation (in the absence of contraindications contraindication) starting from the transesophageal echocardiography.
7. Electrical cardioversion or use of amiodarone, other antiarrhythmic, or drug inducing bradycardia (beta-blockers, bradycardic calcium channel blocker, digitalis, flécaïnamide) in the previous 6 hours before inclusion
8. Contraindication to amiodarone: history of serious adverse event related to amiodarone, history of lung disease related to amiodarone, history of hyperthyroidism related to amiodarone, PR interval > 240 ms, severe sinus node dysfunction with no pacemaker, 2°/ 3° atrioventricular block with no pacemaker, QTc>480 ms, known or treated hyperthyroidism, hypersensitivity to iodine, amiodarone or to any of the excipients, severe hepatocellular insufficiency (prothrombin rate <20%), diffuse Interstitial Lung Disease.
9. Kalemia < 3 mmol/L
10. Pregnant or breast feeding women
11. Moribund patient or death expected from underlying disease during the current admission; Patient deprived of liberty and persons subject to institutional psychiatric care
12. Participation to another interventional trial on septic shock and/or arrhythmic disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 240 (Estimated)
Dates: Start 2021-11-09 (Actual); Primary Completion 2026-02 (Estimated); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
all-cause mortality (a hierarchical criterion) | 28 days
  The duration of septic shock is defined as the time (number of days) from randomization to successful weaning of vasopressors
  The Finkelstein-Schoenfeld method is based on the principle that each patient in the clinical trial is compared with every other patient within each stratum in a pairwise manner. The pairwise comparison proceeds in hierarchical fashion, using all-cause mortality, followed by the duration of septic shock when patients cannot be differentiated on the basis of mortality. This method gives a higher importance to all-cause mortality.
the duration of septic shock according to the Finkelstein-Schoenfeld method (a hierarchical criterion). | 28 days
  The duration of septic shock is defined as the time (number of days) from randomization to successful weaning of vasopressors
  The Finkelstein-Schoenfeld method is based on the principle that each patient in the clinical trial is compared with every other patient within each stratum in a pairwise manner. The pairwise comparison proceeds in hierarchical fashion, using all-cause mortality, followed by the duration of septic shock when patients cannot be differentiated on the basis of mortality. This method gives a higher importance to all-cause mortality.

SECONDARY OUTCOMES:
Rhythm efficacy at day-7 (or at discharge or death if before day-7) | up to 7 days
  1. Number of patients with sinus rhythm
  2. Number of days alive with sinus rhythm
  3. Number of days alive with NOSVA and heart rate < 110 bpm
  4. Proportion of patients receiving therapeutic anticoagulation after randomisation
Morbimortality | Day 28
  1. Duration of septic shock and Length of stay in intensive care unit and in hospital at day-28
  2. Proportion of patients alive free from vasopressors at day-7 (or at discharge or death if before day-7)
  3. Arterial lactate clearance at day-3 defined as the percentage of arterial lactate decrease between lactate at randomisation (day-1) and at day-3.
  4. Proportion of patients alive free from organ dysfunction at day-7 (or at discharge or death if before day-7)
  5. All-cause deaths at day-28.
Tolerance at day-7 and day-28 | Day 7 and day 28
  1. Proportion of patients with at least one arterial thrombotic event including ischemic stroke and non-cerebrovascular arterial thrombotic event
  2. Proportion of patients with at least one major bleeding event according to the International Society of Thrombosis and Haemostasis definition at Day-28;
  3. Proportion of patients with at least one serious adverse event related to amiodarone or to magnesium sulfate; and proportion of each type of event
  4. Proportion of patients presenting at least one serious adverse event associated with electrical cardioversion (for patients receiving electrical cardioversion).

CONTACTS AND LOCATIONS:
Overall Officials: Vincent LABBE, MD, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (1):
- Service de Médecine Intensive Réanimation-Hôpital Tenon, Paris, France

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Labbe V, Desnos C, Preau S, Doyen D, Contou D, Bagate F, Souweine B, Pey V, Bertrand PM, Muller G, Boissier F, Asfar P, Bonnet N, Joffre J, Sy O, Dres M, Annoni F, Monnet X, Carreira S, Vivier E, Serck N, Wiart A, Voicu S, Heming N, Le Breton C, Chevrel G, Chemouni F, Piagnerelli M, Haentjens L, Fartoukh M, Taccone F, Durand D, Monthieux G, Berard L, Rousseau A, Mekontso Dessap A. Risk, rate or rhythm control for new onset supraventricular arrhythmia during septic shock: protocol for the CAFS multicentre, parallel-group, open-label trial. BMJ Open. 2025 Apr 1;15(4):e090404. doi: 10.1136/bmjopen-2024-090404. PMID 40169282